CLINICAL TRIAL: NCT01348659
Title: Effects of Hypertonic Saline-hydroxyethyl Starch Solution on Extracellular Water in Cardiac Surgery Patients
Brief Title: Effects of Hypertonic Saline-HES Solution on Extracellular Water in Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kati Järvelä (Other)
Collaborators: Finnish Cultural Foundation (Other)
Responsible Party: Sponsor-Investigator, Kati Järvelä, MD, PhD, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R09246M; 2010-019352-42 (EudraCT Number)
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Fluid Volume Disorder
Keywords: Hypertonic saline; Extracellular fluid; cardiopulmonary bypass
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7.2% NaCl/hydroxyethyl starch (Active Comparator): 250 ml of 7.2% NaCl in hydroxyethylstarch (HES 200/0,5) (Hyperhaes®, Fresenius Kabi)
  Interventions: Drug: 7.2% NaCl/hydroxyethylstarch
- 0.9% NaCl (Active Comparator): 250 ml of NaCl 0.9% (Natriumklorid Braun 9 mg/ml)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: 7.2% NaCl/hydroxyethylstarch — 250 ml of 7.2% NaCl in hydroxyethylstarch (HES 200/0,5) will be given into the venous reservoir of the cardiopulmonary bypass circuit after aortic declamping.
  Other Names: Hyperhaes®, Fresenius Kabi
  Arms: 7.2% NaCl/hydroxyethyl starch
Drug: NaCl 0.9% — 250 ml of NaCl 0.9% will be given into the venous reservoir of the CPB circuit after aortic declamping.
  Other Names: Natriumklorid Braun 9 mg/ml
  Arms: 0.9% NaCl

SUMMARY:
The aim of the study is to describe the effects of hypertonic saline/hydroxyethylstarch solution in comparison to saline solution for 25 + 25 patients undergoing coronary bypass grafting surgery (CABG) using CPB. The study fluid will be given into the venous reservoir of the CPB circuit after aortic declamping. Primary endpoints are the changes in body weight and extracellular water from baseline to the first postoperative morning.

DETAILED DESCRIPTION:
Cardiac surgery and cardiopulmonary bypass (CPB) cause fluid retention in the body. Both dilution of serum proteins and destruction of vascular endothelial glycocalyx cause extravasation of the fluids. We cannot avoid this phenomenon but we can try to restore the excess fluid into the intravascular space where it can be excreted via the kidneys.

Hypertonic saline (HS) creates an osmotic gradient across the cellular membrane, causing a fluid shift from the intracellular space into the extracellular space and from the extravascular space into the intravascular space. The intravascular hypertonic benefit is short-lasting as a result of redistribution of fluid between the intravascular and interstitial spaces. The effect can be lengthened by adding colloid component into the solution.

The aim of the study is to describe the effects of hypertonic saline/hydroxyethylstarch solution in comparison to saline solution for 25 + 25 patients undergoing coronary bypass grafting surgery (CABG) using CPB. The study fluid will be given into the venous reservoir of the CPB circuit after aortic declamping. Primary endpoints are the changes in body weight and extracellular water from baseline to the first postoperative morning. Secondary endpoints are the need of fluids and diuretic medication during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* male gender and no need for pulmonary artery catheter (pulmonary hypertension or left ventricular ejection fraction < 40%).

Exclusion Criteria:

* chronic hyponatremia and significant renal dysfunction.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in extracellular water from baseline to the first postoperative morning. | 24h
  Perioperative fluid balance will be assessed by measuring changes in body weight and extracellular water from baseline to the first postoperative morning.

SECONDARY OUTCOMES:
Need of fluids during the day of surgery. | 24h
  Need of fluids and diuretic medication during the day of surgery until the first postoperative morning will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kati Järvelä, MD, PhD, Principal Investigator — Tampere University Hospital Heart Center
Locations (1):
- Tampere University Hospital Heart Center, Tampere, Finland